CLINICAL TRIAL: NCT06281249
Title: Real-time Spine Ultrasound Imaging System: Data Collection Study
Brief Title: Neuraxial Ultrasound Device Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Rivanna Medical, Inc. (Unknown)
Responsible Party: Principal Investigator, Clemens Ortner, Clinical Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 73172
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Labor Pain; Cesarean Delivery Regional Anesthesia Induction
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Intrathecal neuraxial procedure (Experimental): Participants undergoing surgery, receiving neuraxial intrathecal anesthesia with block placement in part by the investigational device.
  Interventions: Device: Ultrasound placement device

INTERVENTIONS:
Device: Ultrasound placement device — Device to assist in placement of epidural procedure
  Other Names: Accuro 3S

SUMMARY:
The aim of the study is to develop a device that can eliminate failed neuraxial placements in challenging patients.The study will attempt to improve safety and efficacy of neuraxial anesthesia with high precision real-time needle visualization through automated real-time needle guidance at the bedside with an experimental device (Accuro 3S). Investigators will verify the clinical workflow for utilizing the Accuro 3S during epidural and spinal procedures and validation of needle visualization while using the device as well as anatomical guidance provided by the device during spinal imaging.The underlying bone imaging enhancement algorithms were introduced in the commercially available FDA approved Accuro. The Accuro 3S will be used to establish needle insertion point and trajectory, after which the clinician will use standard of care methods to advance the needle such as the loss of resistance method.

DETAILED DESCRIPTION:
This is a prospective, structured observational study (data collection study) in which Investigators enroll patients who are scheduled for neuraxial anesthesia procedures.

Qualified subjects will be identified and contacted by the anesthesia team prior to their clinical evaluation for labor neuraxial analgesia. Potential patients will be informed of the study, and if study individuals choose to participate and an informed consent form will be signed prior to any study related activities.

When study participants request labor analgesia, investigators will incorporate routine care delivery flow for patients receiving ultrasound guided neuraxial anesthesia.

The clinician will apply ultrasound gel to the Accuro 3S probe (gel inside the probe need not be sterile), and then cover the probe in a sterile probe cover. Sterile ultrasound gel will then be applied to the patient's skin on the back to enable imaging. The Accuro 3S probe will be applied to the patient's spinal region and the clinician will perform scouting scans. Image recordings can be captured by depressing a button located on the probe handle. While performing the scouting scans, the provider will take several image recordings of the spine. The image recordings will include two levels, finding the space, and then at each level plus a spinous process, scanning left and right at each of these points.

The clinician will then administer local anesthetic prior to needle procedures. After needle insertion point and trajectory is established on the ultrasound image, the epidural or spinal needle will then be advanced by the clinician based on their standard technique. While advancing the needle the provider will collect a series of image recordings.

After proper placement of needle/catheter, the Accuro 3S device will then be removed from the patient and they will proceed with standard clinical protocol for post placement care.

Accuro 3S: Primary data collected during this study will be images recordings captured during the scouting and needle placement for the epidural procedure. Images will be acquired directly on the 3S and will not contain patient identifiers.

After collection of data up to 100 patients, Investigators will be moving to clinical analysis.

Rivanna is the sponsor and will be funding this research. The de-identified patient data that Rivanna will receive for analysis include: results of demographic information (e.g. age, height, weight, sex, race, and ethnicity). Obstetric details including gravity, parity, gestational age, labor or cesarean delivery, pain score prior to and after placement. Accuro 3S Images (including scouting images of spine and images of needle placement). Insertion: Number of needle passes and redirects, interspace attempted/inserted; epidural or spinal, and needle gauges used. Number, type, and details of any complication (e.g. wet tap). Failed spinal or epidural including: pain >3/10 after labor epidural, catheter replacement, no or one-sided sensory block, failure to provide cesarean anesthesia, conversion to different type of anesthesia.

Patients will undergo their standard medical and obstetric treatment at the discretion of the obstetrical and anesthesia team. There will be no delay in their treatment due to this study, and the device data will not be available of influence care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* The patient is eligible for placement of neuraxial anesthesia, and the patient has agreed to the procedure.
* Patient skin is intact in the area of placement of the epidural or spinal anesthesia.

Exclusion Criteria:

* Contraindication to epidural catheter placement including bleeding diathesis (essential thrombocythemia, idiopathic thrombocytopenic purpura, von Willebrand disease, and hemophilia A or B), neurological dysfunction (multiple sclerosis, subacute myeloopticoneuropathy or preexisting lower limb neurological deficit), prior extensive spinal surgery or major spinal deformity, pre-operative use of anti-coagulant with planned use of therapeutic dose of anti-coagulant in post-operatively, documented pre-operative coagulopathy (INR greater than 1.3 not on Coumadin or PTT greater than 42), platelets less than 70,000/μL, or evidence of infection at potential epidural site.
* Presence of orthopedic implants in the spine.
* Skin dyscrasias or allergies to the ultrasound procedure.
* Unable to assume sitting position.
* Body Mass Index (BMI) less than 20 kg/m2.
* Known allergies to ultrasound gel.
* Known history of allergic reactions to adhesives used in standard epidural placement

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of difficult block placement | 15 minutes
  Difficult block placement is defined by need of > 2 needle insertion attempts for succesful neuraxial analgesia/anesthesia

SECONDARY OUTCOMES:
Incidence of failed block | 30 minutes
  Failed labor epidural analgesia and spinal anesthesia will be defined by presence of 1 or more of the following conditions: one-sided or no sensory block, pain >3/10 after epidural placement, epidural replacement, conversion to a different form of anesthesia)
Incidence of post-dural puncture headache | 7 days
  Headache developing within 7 days post block placement defined by presence of at least one of the following symptoms: posture dependent headache, symmetric headache posture dependent, neck pain posture dependent

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Ortner, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boselli E, Hopkins P, Lamperti M, Estebe JP, Fuzier R, Biasucci DG, Disma N, Pittiruti M, Traskaite V, Macas A, Breschan C, Vailati D, Subert M. European Society of Anaesthesiology and Intensive Care Guidelines on peri-operative use of ultrasound for regional anaesthesia (PERSEUS regional anesthesia): Peripheral nerves blocks and neuraxial anaesthesia. Eur J Anaesthesiol. 2021 Mar 1;38(3):219-250. doi: 10.1097/EJA.0000000000001383. PMID 33186303
- [Background] Practice Guidelines for Obstetric Anesthesia: An Updated Report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia and the Society for Obstetric Anesthesia and Perinatology. Anesthesiology. 2016 Feb;124(2):270-300. doi: 10.1097/ALN.0000000000000935. No abstract available. PMID 26580836
- [Background] Ring L, Landau R, Delgado C. The Current Role of General Anesthesia for Cesarean Delivery. Curr Anesthesiol Rep. 2021;11(1):18-27. doi: 10.1007/s40140-021-00437-6. Epub 2021 Feb 24. PMID 33642943
- [Background] Rajagopalan S, Shah K, Guffey D, Tran C, Suresh M, Wali A. Predictors of difficult epidural placement in pregnant women: A trainees' perspective. J Anaesthesiol Clin Pharmacol. 2019 Oct-Dec;35(4):548-552. doi: 10.4103/joacp.JOACP_340_18. PMID 31920244
- [Background] Ismail S, Raza A, Munshi K, Tabassum R. Failure rate of labor epidural: An observational study among different levels of trainee anesthesiologists in a university hospital of a developing country. J Anaesthesiol Clin Pharmacol. 2021 Apr-Jun;37(2):210-215. doi: 10.4103/joacp.JOACP_39_19. Epub 2021 Jul 15. PMID 34349368
- [Background] Cittadini G, Martinoli C. [Ultrasound and the bone: a difficult relationship]. Radiol Med. 1995 Jan-Feb;89(1-2):12-7. Italian. PMID 7716291
- [Background] Mao Q, He H, Lu Y, Hu Y, Wang Z, Gan M, Yan H, Chen L. Ultrasound probe tilt impedes the needle-beam alignment during the ultrasound-guided procedures. Sci Rep. 2021 Jan 15;11(1):1599. doi: 10.1038/s41598-021-81354-w. PMID 33452406
- [Background] Tiouririne M, Dixon AJ, Mauldin FW Jr, Scalzo D, Krishnaraj A. Imaging Performance of a Handheld Ultrasound System With Real-Time Computer-Aided Detection of Lumbar Spine Anatomy: A Feasibility Study. Invest Radiol. 2017 Aug;52(8):447-455. doi: 10.1097/RLI.0000000000000361. PMID 28230717